CLINICAL TRIAL: NCT06145776
Title: Effects of Cognitive-motor Dual-Task Training and tDCS on Brain Electrical Activity Assessed by EEG and Cognitive Performance in Patients With Parkinson's Disease: a Randomized, Double-blind, Controlled Clinical Trial.
Brief Title: The Role of EEG in Identifying Cognitive Changes in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Suellen Andrade, Suellen Marinho Andrade, Federal University of Paraíba, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EEG_DPcog
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease; Cognition Disorder; EEG With Abnormally Slow Frequencies
Keywords: Parkinson; EEG; cognition; dual-task cost
MeSH Terms: conditions — Parkinson Disease; Cognition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, group controlled clinical trial. Parallel study,
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly allocated, using an online generator (www.random.org), into two groups (1:1): CG) tDCS active + gait training; EG) tDCS active + gait training + dual-task. This sequence will be performed independently and remotely by a blinded investigator, who will have no knowledge of other study procedures. The concealed allocation process will be conducted using sequentially numbered sealed opaque envelopes. The outcome assessors and patients will be blinded to the procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dual-task group (Experimental): Dual-Task Training Protocol (DTTP) The dual-task training protocol (DT) will consist in cognitive exercise categories: verbal fluency, mental screening tasks, discrimination, decision-making and reaction time tasks, which will be associated to treadmill gait training (Sousa et al., 2016). Verbal commands will focus on the following: (1) large strides; (2) heel strike; (3) raising the knees while walking (Kelly et al., 2012).
  Interventions: Other: tDCS + tredmill training (Standart trehab training); Other: Cognitite-motor Dual Task Training (DT training)
- control group (Active Comparator): The participants will perform 21 min treadmill gait training associated to tDCS active in F3 for 20 min, 3 times a week for 4 weeks.
  Interventions: Other: tDCS + tredmill training (Standart trehab training)

INTERVENTIONS:
Other: tDCS + tredmill training (Standart trehab training) — Standart Rehab training will consist in 20 min treadmill gait training associated to active atDCS F3 2mA for 20 min.
Other: Cognitite-motor Dual Task Training (DT training) — The dual-task training protocol (DT) will consist in cognitive exercises (verbal fluency, mental screening tasks, discrimination, decision-making and reaction time tasks) and motor exercises (walking while carrying a tray with only one empty glasscarrying a glass while walks, change peaces from one pocket to another, looking from one side to another while walking)
  Arms: dual-task group

SUMMARY:
This study is a group controlled clinical trial. Parallel study, patients aged 40-80 years, with Parkinson disease. Twelve sessions, three times a week, for 30 minutes. Training will consist of Transcranial Direct Current Stimulation linked to tredmill training, in 3 blocks of 7 minutes, and adicionally to the Experimental Group, dual-task cognitive-motor exercises, simultaneously. The investigators will use the folowwing instruments: Auditory Stroop Test, Trail Making Test, Montreal Cognitive Assessment, Timed-up-and-go ST and DT, UPDRS II and III and Eletroencefalography (EEG). The objective is to examine cognitive alterations on PD pacients due to intervention and the relationships between baseline outcomes in responders and non-responders to therapy.

DETAILED DESCRIPTION:
Background: Parkinson disease (PD) is one of the most common age-related brain disorders. PD is defined primarily as a movement disorder, with the typical symptoms being resting tremor, rigidity, bradykinesia and postural instability. In addition to the defining dopamine-related motor symptoms, however, PD is increasingly recognized as a heterogeneous multisystem disorder involving other neurotransmitter systems, such as the serotonergic, noradrenergic and cholinergic circuits. Thus, a wide variety of nonmotor symptoms (NMS) linked with these neurotransmitters are commonly observed in patients with PD. Cognitive decline is among the most common and important NMS. Robust evidence indicates that in comparison with age-matched groups without PD, people with PD exhibit more rapid decline in a number of cognitive domains - in particular, executive, attentional and visuospatial domains, but also memory. In recent years, research has focused on the pre-dementia stages of cognitive impairment in PD, including mild cognitive impairment (MCI). Several longitudinal studies have shown that MCI is a harbinger of dementia in PD, although the course is variable, and stabilization of cognition - or even reversal to normal cognition - is not uncommon. A variety of biomarkers have been studied, some using novel structural and functional imaging techniques, and have documented in vivo brain changes associated with cognitive impairment. Patients with Parkinson's disease have difficulty performing a dual-task, a condition present in everyday life. It is possible that strategies such as Transcranial Direct Current Stimulation can be associated with motor training enriched with dual-task and cognitive training to improve the performance of two concurrent tasks. It is currently unclear whether specific tasks and clinical conditions of PD patients have different results after the intervention. Therefore, the proposed randomized controlled trial will examine the effects of a intervention protocol on brain eletric activity and cognitive outcomes on PD patientes and the relationships between baseline outcomes in responders and non-responders to therapy.

Discussion: This study will evaluate the effectiveness of an intervention protocol with transcranial direct current stimulation, dual-task motor-cognitive training in patients with Parkinson's disease. The study will also highlight whether, by qEEG analysis, the clinical factors and variability between individuals that could interfere in the efficacy intervention and influence the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with idiopathic Parkinson's disease by a neurologist based on definitive evidence of responsiveness to levodopa at the start of the disease and the history of progressive hypokinesia with asymmetric onset. PD will be diagnosed based on Parkinson's Disease Society Brain Bank (PDSBB) criteria, as described in Hughes et al. (1992)
* Age between 40 and 70 years, with no distinction for sex, schooling level or other sociodemographic characteristics;
* disease staging between 1.5 and 3, according to the modified Hoehn and Yahr scale (Hoehn and Yahr, 1998);
* undergoing regular pharmacological treatment with levodopa (equivalent dose > 300 mg) or taking antiparkinsonian medication, such as anticholinergics, selegiline, dopamine agonists, and COMT (catechol-O-methyl transferase) inhibitors for at least 4 weeks prior intervention;
* score of more than 24 points on the Mini-Mental State Examination (Folstein et al., 1975);
* not exhibiting other associated neurological diseases; and
* no musculoskeletal and/or cardiorespiratory changes that could compromise gait.

Exclusion Criteria:

* diagnosis of atypical Parkinson's disease;
* neuropsychiatric comorbidities;
* convulsions, metal clips and/or pacemaker;
* deep brain stimulation implant;
* history of epilepsy; neurosurgery;
* traumatic brain injury;
* alcohol abuse or drug dependency;
* associated diseases of the peripheral or central nervous system;
* undergoing physical therapy at another location;
* inability to walk 10 meters;
* presence of important dyskinesia that prevents the participant from sitting in a chair;
* abnormal and persistent increase in systemic blood pressure before or during training, after three measurements taken 5 min apart-Cut-off: systolic blood pressure ≥ 140 mm Hg and/or diastolic ≥ 90 mm Hg (Malachias et al., 2016);
* not understanding any of the training protocol stages; chemical scalp treatment within the previous 30 days, and experiencing severe pain and/or discomfort that precludes performing the proposed activities.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
EEG outcomes | 30 days
  PSD of theta, alpha and beta and alpha/theta ratio and beta/theta ratio of 6 ROIs (righ and left: frontal, temporoparietal and occipital)
clinic outcome | 30 days
  Dual-task cost

SECONDARY OUTCOMES:
Total Montreal Cognitive Assessment (MoCA) | 30 days
  total score obtained at Montreal Cognitive Assesment, for a possible maximum of 30 points. A final total score of 26 and above is considered normal.
domains of MoCA | 30 days
  Score of ecah subscale obtained at Montreal Cognitive Assesment: visuospatial/executive (5 points); nomination (3 points); memory (5 points for delayed recall); attention (6 points); language (3 points); abstraction (2 points); and orientation (6 points).
Trail Making Test part B (TMT-B) | 30 days
  TMT-B is scored based on how long it takes to complete the test, within 5 minutes.
Stroop Test | 30 days
  score of total Stroop test (Stroop Colors and Stroop Words). Word, color, and color-word T-Scores of 40 or less are considered "low." Word, color, and color-word T-Scores above 40 or are considered "normal."
Movement Disorder Society - Unified Parkinson's Disease Rating Scale PART II Score Compare insights MDS-Unified Parkinson's Disease Rating Scale part II (UPDRS-II) | 30 days
  Score of part II of UPDRS, Motor experiences of daily living: 13 items. Score range: 0-52,[8] 12 and below is mild, 30 and above is severe

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, Doctor, Principal Investigator — Federal University of Paraiba
Locations (2):
- Brazil (2):
  - Federal University of Paraiba, João Pessoa, Paraíba
  - Aging and Neuroscience Studies Laboratory, João Pessoa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costa-Ribeiro A, Andrade SMMDS, Ferrer MLV, Silva OAPD, Salvador MLS, Smaili S, Lindquist ARR. Can Task Specificity Impact tDCS-Linked to Dual Task Training Gains in Parkinson's Disease? A Protocol for a Randomized Controlled Trial. Front Aging Neurosci. 2021 Jul 1;13:684689. doi: 10.3389/fnagi.2021.684689. eCollection 2021. PMID 34276344